CLINICAL TRIAL: NCT07029386
Title: The Effectiveness of Individualized Transcranial Electrical Stimulation in Improving Cognitive Impairment in Patients With Central Nervous System Inflammatory Demyelinating Diseases
Brief Title: Effects of Transcranial Electrical Stimulation on Cognitive Impairment in CNS Inflammatory Demyelinating Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: xw-tES-01
Record Dates: First submitted 2025-01-19; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Idiopathic Inflammatory Demyelinating Disorders of the Central Nervous System

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromodulation Group (Active Comparator)
  Interventions: Device: tES
- sham Neuromodulation Group (Sham Comparator)
  Interventions: Device: tES

INTERVENTIONS:
Device: tES — his study employs a randomized controlled trial (RCT) design, randomly dividing eligible participants into a neuromodulation group and a sham neuromodulation group.
  Neuromodulation Group:
  Receive individualized transcranial electrical stimulation (tES) treatment Combined with cognitive training
  Stimulation parameters:
  Total current: approximately 2mA Duration: 21 minutes Electroencephalogram (EEG) and functional MRI (fMRI) monitoring before and after electrical stimulation
  Arms: Neuromodulation Group
Device: tES — Use the same device and procedure as the neuromodulation group Stimulation device automatically turns off after 30 seconds Maintain device connection Design creates similar initial sensations to actual stimulation Maintains the double-blind nature of the study
  Arms: sham Neuromodulation Group

SUMMARY:
Background: Central nervous system inflammatory demyelinating diseases often lead to significant cognitive impairment, presenting a critical challenge in patient management.

Objective: To evaluate the effectiveness of individualized transcranial electrical stimulation (tES) in improving cognitive function among patients with inflammatory demyelinating disorders.

Methods: This study will assess cognitive performance through standardized neuropsychological assessments before and after individualized tES intervention, measuring changes in cognitive domains including memory, attention, executive function, and processing speed.

Anticipated Results: the investigators hypothesize that personalized transcranial electrical stimulation will demonstrate significant improvements in cognitive performance, potentially offering a non-invasive therapeutic approach for managing cognitive decline in central nervous system inflammatory demyelinating diseases.

Significance: This research may provide novel insights into neuromodulation strategies for cognitive rehabilitation in patients with complex neurological conditions.

ELIGIBILITY:
Inclusion Criteria:、

1. Patients with Neuromyelitis Optica Spectrum Disorders (NMOSD), Multiple Sclerosis (MS), and other Central Nervous System Inflammatory Demyelinating Diseases that meet diagnostic criteria;
2. Patients with SDMT scores <55 or subjective cognitive decline;
3. Age between 18 and 65 years, gender unrestricted;
4. Hamilton Anxiety and Depression Scale scores <7 points for both scales;
5. No relapse or medication changes in the past month;
6. EDSS (Expanded Disability Status Scale) score ≤6;
7. Right-handed, native Chinese speakers with sufficient educational background to understand the test instructions;
8. Willing to participate and have signed informed consent.-

Exclusion Criteria:

1. Relapse record within the past month;
2. Medication adjustment within the past month or having undergone modified electroconvulsive therapy, transcranial magnetic stimulation, or other neuromodulation techniques;
3. Participating in any other clinical research within 1 month prior to enrollment or currently;
4. Presence of cochlear hearing aids, cardiac pacemakers, or implanted brain stimulation devices;
5. Skin integrity damage at electrode placement sites, or allergy to electrode gel or adhesives;
6. History of epilepsy, hydrocephalus, central nervous system tumors, brain injury, or intracranial infections;
7. Pregnant or lactating women, or those planning pregnancy in the near future;
8. Scoring ≥3 on item 3 (suicide item) of the HDRS-17 or concurrent severe mental illness;
9. Concurrent severe or unstable organic diseases;
10. Unable to cooperate with treatment, follow-up, or clinical, EEG, and imaging data collection due to poor patient compliance;
11. Other situations deemed inappropriate for study participation by the researchers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive Assessments | Before treatment, on the last 1 day of treatment, and one month after treatment.
  AVLT, Auditory Verbal Learning Test AVLT score is higher, the better.

SECONDARY OUTCOMES:
SDMT | Before treatment, on the last 1 day of treatment, and one month after treatment
  symbol digit modalities test, SDMT score is higher, the better."
Improvement in EEG Parameters | Before treatment, on the last 1 day of treatment, and one month after treatment
  the power spectral density (PSD) of delta, theta, alpha, beta, and gamma waves; t Default Mode Network (DMN), Sensory Motor Network (SMN), Visual Network (VN), Auditory Network (AN), Cognitive Control Network (CCN), Salience Network (SN), and Dorsal Attention Network (DAN); the intranetwork connectivity within these networks; and the internetwork connectivity between these networks.
Improvement in fMRI Parameters | Before treatment, on the last 1 day of treatment, and one month after treatment
  Default Mode Network (DMN), Sensory Motor Network (SMN), Visual Network (VN), Auditory Network (AN), Cognitive Control Network (CCN), Salience Network (SN), and Dorsal Attention Network (DAN); the intranetwork connectivity within these networks; and the internetwork connectivity between these networks.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No